CLINICAL TRIAL: NCT06706271
Title: The Effect of Vitamin D3 Supplementation on Hepcidin and Ferritin Serum Levels in Children With Chronic Kidney Disease
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Hasanuddin University (Other)
Responsible Party: Principal Investigator, Andi Muldiana Dwi Rachmayani, Pediatric Resident, Department of Pediatric, Hasanuddin University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C105201005
Record Dates: First submitted 2024-11-23; First posted 2024-11-26 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Chronic Kidney Disease Stage 1; Chronic Kidney Disease Stage 2
Keywords: Chronic Kidney Disease; Vitamin D; Hepcidin; Ferritin; Vitamin D3
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Vitamin D

STUDY DESIGN:
Intervention Model Description: The study targets children diagnosed with chronic kidney disease, categorized into two groups based on their glomerular filtration rate (GFR): those with GFR < 90 mL/min/1.73 m² and those with GFR ≥ 90 mL/min/1.73 m². Participants are selected through purposive sampling, ensuring they meet defined inclusion criteria related to age, CKD diagnosis, and baseline serum levels. Serum levels of vitamin D, hepcidin, and ferritin are measured before and after vitamin D3 supplementation. This allows for comparative analysis of changes within each group and between the two groups, providing insights into the effects of vitamin D3 on iron metabolism.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- GFR more than 90 mL/min/1,73 m2 (Experimental): Children with GFR more than 90 mL/min/1,73 m2, and will be given 2000 IU of Vitamin D for 6 weeks
  Interventions: Drug: Vitamin D
- GFR less than 90 mL/min/1,73 m2 (Experimental): Children with GFR less than 90 mL/min/1,73 m2, and will be given 2000 IU of Vitamin D for 6 weeks
  Interventions: Drug: Vitamin D

INTERVENTIONS:
Drug: Vitamin D — 2000 IU of Vitamin D

SUMMARY:
The goal of this clinical trial is to analyze the effects of in vitamin D3 on serum hepcidin and ferritin levels among children with chronic kidney disease. The main questions it aims to answer is:

"What is the effect of giving vitamin D3 on serum hepcidin and ferritin levels in children with chronic kidney disease?"

We will compare the effect of vitamin D3 administration on hepcidin and ferritin between 2 groups. Group A consists of children with GFR more 90 mL/min/1,73 m2. Group B consists of children with GFR less than 90 mL/min/1,73 m2

Participants will be given the same 2000 IU of Vitamin D/day for 6 weeks.

DETAILED DESCRIPTION:
The primary objective of the study is to analyze the effects of vitamin D3 administration on serum levels of hepcidin and ferritin in children diagnosed with CKD. The research aims to measure these serum levels before and after vitamin D3 supplementation across different stages of kidney function, categorized by glomerular filtration rate (GFR). Specifically, it seeks to determine whether vitamin D3 can effectively reduce hepcidin levels and improve iron status as indicated by ferritin levels. The study employs a structured methodology involving children with CKD, divided into two groups based on their GFR: those with GFR < 90 mL/min/1.73 m² and those with GFR ≥ 90 mL/min/1.73 m². Serum levels of vitamin D, hepcidin, and ferritin will be measured at baseline (before supplementation) and after a defined period of vitamin D3 administration. The research will utilize statistical analyses to compare these values within and between groups to establish any significant changes attributable to the supplementation.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 2 to 18 years diagnosed with chronic kidney diseases at Dr. Wahidin Sudirohusodo hospital
* Parents have signed their child's consent to participate in the study

Exclusion Criteria:

* History of blood transfusion 3 months prior
* Liver dysfunction
* Sepsis
* Routine consumption of Vitamin D
* Routine consumption of iron supplement
* Patients diagnosed with iron deficiency anemia

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 43 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-09-02 (Actual)

PRIMARY OUTCOMES:
Vitamin D Level | From enrollment to the end of treatment at 6 weeks
  Vitamin D is measured before and after supplementation of Vitamin D
Ferritin Level | From enrollment to the end of treatment at 6 weeks
  Ferritin level before and after Vitamin D supplementation
Hepcidin level | From enrollment to the end of treatment at 6 weeks
  Hepcidin level before and after Vitamin D supplementation

CONTACTS AND LOCATIONS:
Overall Officials: Andi Muldiana Dwi Rachmayani, MD, Principal Investigator — Hasanuddin University
Locations (1):
- Wahidin Sudirohusodo Hospital, Makassar, South Sulawesi, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Altemose KE, Kumar J, Portale AA, Warady BA, Furth SL, Fadrowski JJ, Atkinson MA. Vitamin D insufficiency, hemoglobin, and anemia in children with chronic kidney disease. Pediatr Nephrol. 2018 Nov;33(11):2131-2136. doi: 10.1007/s00467-018-4020-5. Epub 2018 Jul 14. PMID 30008129
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/30008129/

DOCUMENTS (1):
  • Study Protocol (2023-05-01): https://cdn.clinicaltrials.gov/large-docs/71/NCT06706271/Prot_000.pdf